CLINICAL TRIAL: NCT00798902
Title: A Multi-Center, Prospective, Parallel Group, Randomized, Pilot Study Evaluating Safety and Preliminary Effectiveness Of Prefix Compared To Iliac Crest Bone In Subjects With DDD Undergoing Transforaminal Lumbar Interbody Fusion
Brief Title: Pilot Study to Assess Safety/Preliminary Effectiveness of Prefix in Subjects With Degenerative Disc Disease (DDD) Undergoing Spine Fusion Surgery
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: BioSurface Engineering Technologies, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PFX-100
Record Dates: First submitted 2008-11-24; First posted 2008-11-26 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Degenerative Disc Disease; Spondylolisthesis
Keywords: DDD; Spondylolisthesis; Spine Fusion; Lumbar Spine; Bone Graft
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spondylolisthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): Iliac Crest Autograft
  Interventions: Other: Iliac crest autograft
- Prefix 150 (Experimental): Prefix (AMPLEX) B2A Peptide Enhanced Ceramic Granules
  Interventions: Device: Prefix (AMPLEX) B2A Peptide Enhanced Ceramic Granules

INTERVENTIONS:
Device: Prefix (AMPLEX) B2A Peptide Enhanced Ceramic Granules — 150 micrograms/cc BVF
  Other Names: AMPLEX
  Arms: Prefix 150
Other: Iliac crest autograft — autograft
  Arms: Control

SUMMARY:
This is a pilot study to evaulate the safety and prelimary effectiveness of Prefix as compared to autogenous bone for spinal fusion procedures in skeletally mature subjects with degenerative disc disease (DDD) at one level from L2-S1.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of DDD requiring single level fusion (L2-S1) with up to Grade I Spondylolisthesis
* Have a preoperative screening qualifying VAS and ODI scores
* Be a skeletally mature male or a non-pregnant, non-lactating female, age 18 -70 inclusive
* Have not been sufficiently responsive to at least 6 months of non-operative treatment prior to study enrollment

Exclusion Criteria:

* Are female subjects who are pregnant or nursing, or women planning to become pregnant during the first year (12 months) following the surgery
* A history of previous surgery in the lumbar spine with or without attempted fusion
* Grade II or greater spondylolisthesis
* More than 0 degrees of kyphosis at the operated disc space
* Evidence of scoliosis in the lumbar region of more than 10 degrees
* Collapsed disc space with bridging osteophytes
* A systemic or local infection at the site of surgery
* An acute fracture of the spine at the time of enrollment in the study
* An active history of systemic malignancy
* A medical condition, serious intercurrent illness, or extenuating circumstance that, in the opinion of the Investigator, would preclude participation in the study
* A known hypersensitivity to any of the components of the product or a known titanium allergy or a known allergy to polyetheretherketone (PEEK)
* A history of any autoimmune disease, such as, systemic lupus erythematosus, Addison's disease, Crohn's disease, or rheumatoid arthritis
* A history of any severe allergy or anaphylaxis, or a history of hypersensitivity to protein pharmaceuticals, or have had any previous exposure to a protein pharmaceutical
* Are receiving treatment (before or during surgery) with a drug (e.g., steroids, methotrexate, etc.) that interferes with bone metabolism or are being treated with a bone growth stimulator
* A medical condition requiring radiation, chemotherapy or immunosuppression, or a medical condition requiring systemic corticosteroids
* Are covered under workmen's compensation insurance or prisoners
* Are transient or have been treated in the last 6 months before enrollment for alcohol and/or drug abuse in an in-subject substance abuse program
* Have participated in clinical studies within 3 months of enrollment
* Have a body mass index (BMI) greater than 35
* Use tobacco products (also includes, e.g. nicotine patch or nicotine gum), or have smoked cigarettes within 6 weeks preceding enrollment
* Known to require additional surgery to the lumbar spinal region within the next 6 months
* Have symptomatic multilevel degenerative disease requiring possible instrumented fusion of more than one vertebral level
* Have previously been treated with, or exposed to, therapeutic levels of Bone Morphogenetic Proteins (BMPs), i.e., synthetic or recombinant
* Have a documented medical history or radiographic evidence of a metabolic bone disease (e.g., osteoporosis or osteopenia) or other condition which would negatively impact the bone healing process (e.g. history of Paget's disease, osteomalacia, or other osteodystrophy) or preclude the subject from receiving pedicle screw fixation
* Are involved in or planning to engage in litigation related to back and/or leg pain
* Require chronic SQ or IV heparin therapies
* Have an Osteoporosis Risk Assessment Instrument (ORAI) score > to 9 points and, if so, will require a qualifying DEXA scan T score

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2008-11; Primary Completion 2012-07 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Removal/revision or supplemental fixation of the graft material requiring reoperation at the index level, Safety (adverse events), Fusion "success" based on X-rays, Change from baseline in neurological exam scores and ODI scores | 12 months post surgery

SECONDARY OUTCOMES:
Volume of blood loss/transfused blood during surgery, Blinded independent assessment of fusion by CT and other radiographic assessments, Change from baseline in pain scores using VAS and change from baseline in SF-36 v2™ total and subscale scores | 12 months post surgery

CONTACTS AND LOCATIONS:
Overall Officials: David M Hooper, PhD, Study Director — BioSurface Engineering Technologies, Inc
Locations (6):
- United States (6):
  - Confidential, Durango, Colorado
  - Confidential, Washington D.C., District of Columbia
  - University of Kansas Medical Center, Kansas City, Kansas
  - Confidential, Jefferson City, Missouri
  - Confidential, Johnson City, New York
  - Confidential, Tyler, Texas